CLINICAL TRIAL: NCT05595720
Title: Effect of High Intensity Laser on Hemiplegic Shoulder Dysfunction Double Blinded, Placebo-controlled Trial
Brief Title: Effect of High Intensity Laser on Hemiplegic Shoulder Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Deraya U
Record Dates: First submitted 2022-10-17; First posted 2022-10-27 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Shoulder Dislocation or Subluxation
Keywords: Stroke,; Shoulder dysfunction; High intensity laser
MeSH Terms: conditions — Stroke; Shoulder Dislocation; Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental)
  Interventions: Device: hight intenisty laser
- control group (No Intervention)

INTERVENTIONS:
Device: hight intenisty laser — 7W(LAZR-207)/15W(LAZR-215&115)HIGH POWER LASER THERAPYUNIT WITH 2 WAVELENGTHMODES,COMBINATION(810+980 NM) AND SINGLE(1064 NM)
  Arms: treatment group

SUMMARY:
Hemiplegic shoulder pain (HSP) is a common and disabling complication following a stroke, and it may affect the quality of life. It often occurs following two to three months of stroke. Upper limb impairment is seen in 90% of patients affected by stroke.

Numerous causes have been implicated in developing HSP in stroke. This includes muscle flaccidity around the shoulder joint, shoulder subluxation, shoulder-hand syndrome, increased muscle tone, impingement syndrome, frozen shoulder, brachial plexus injury, and the thalamic syndrome.

Muscle paresis, abnormal muscle tone and loss of proprioception following stroke may render the shoulder complex unstable and therefore prone to misalignment.

In recent years, high-intensity laser therapy (HILT) has been considered as a treatment option for shoulder pain.

HILT increases microcirculation and tissue regeneration and lowers edema, inflammation, and pain with its photomechanical, thermal, electrical, and bio stimulating effects in deep tissues that cannot be reached with LILT.

It has some advantages over LILT, i.e., having higher power, greater tissue penetration capacity to deep tissues, the short emission time, and long rest periods preventing heat accumulation.

In recent studies, effectiveness of HILT has been shown in the treatment of subacromial impingement syndrome, rotator cuff tendinopathy, and frozen shoulder.

ELIGIBILITY:
Inclusion Criteria:

* DISORDER MORE THAN 6 MONTHS
* UNILATERAL
* FIRST TIME

Exclusion Criteria:

* Iinflammatory rheumatic disease,
* cervical radiculopathy,
* diabetes mellitus,
* thyroid disease,
* coronary heart disease,
* cardiac pacemaker,
* neurological disease,
* shoulder surgery, and
* shoulder injection in the last 3 months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
PAIN score | 1 MONTH
  McGill pain questioner scale, scoring from zero to 78 zero is the best score seventy eight is the worst score
FUNCTION | 1 MONTH
  UCLA shoulder score from zero to 35 zero is the worst 35 is the best

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes